CLINICAL TRIAL: NCT05750706
Title: Prospective Observational Study on Incidence of Invasive Fungal Infections Among Patients With Acute Lymphoblastic Leukemia Ph-negative
Brief Title: Incidence of Invasive Fungal Infections Among Patients With Acute Lymphoblastic Leukemia Ph-negative
Acronym: SEIFEM
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Asst Degli Spedali Civili Di Brescia (Other)
Responsible Party: Sponsor
Other Study IDs: 4976
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-02

CONDITIONS: Acute Lymphoblastic Leukemia, Adult; Invasive Fungal Infections
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients without invasive fungal infection: Acute lymphoblastic leukemia, no invasive fungal infection
- Patients with invasive fungal infection: Acute lymphoblastic leukemia, invasive fungal infection
  Interventions: Other: observation of invasive fungal infections

INTERVENTIONS:
Other: observation of invasive fungal infections — observation of invasive fungal infections during chemotherapy
  Groups: Patients with invasive fungal infection

SUMMARY:
The study aims to evaluate incidence of invasive antifungal infections among patients with acute lymphoblastic leukemia Ph negative during the first weeks of treatment

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of acute lymphoblastic leukemia Ph negative
* age more than 18 yo

Exclusion Criteria:

* diagnosis of acute lymphoblastic leukemia Ph positive
* acute lymphoblastic leukemia relapsed/refractory
* lymphoblastic lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with B or T acute lymphoblastic leukemia Ph negative
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of invasive fungal infections | 18 months
  Incidence of invasive fungal infections during first week of chemotherapy

SECONDARY OUTCOMES:
Mortality rate | 30 months
  Mortality rate among patients with invasive fungal infections

CONTACTS AND LOCATIONS:
Overall Officials: Marianna Criscuolo, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided